CLINICAL TRIAL: NCT00000443
Title: Pharmacological Treatment for Alcoholism
Brief Title: Ondansetron Treatment for Alcoholism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAJOH10522
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron

INTERVENTIONS:
Drug: ondansetron (Zofran)

SUMMARY:
The purpose of this study is to: a) evaluate the effectiveness of ondansetron (Zofran) in the treatment of alcohol dependent patients; b) investigate whether early versus late onset alcoholism predicts treatment outcome; and c) determine whether the early and late onset groups respond differently to treatment. Individuals will be "typed" into early onset and late onset alcoholism groups. Individuals will be randomly assigned to a 12-week outpatient treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for alcohol dependence.
* Subjects with early onset alcoholism must also have a diagnosis of antisocial personality disorder.
* Understand the requirements of the study and be able to complete the questionnaires and rating scales.

Exclusion Criteria:

* Current diagnosis of substance dependence or self-report of having used narcotics (opiates, cocaine, amphetamine-like substances, and hallucinogens) in the 30 day period prior to study.
* Positive urine drug screen test for narcotics, barbiturates, or benzodiazepines.
* Receiving current psychotropic medications.
* Current history of other psychiatric disorders excluding nicotine dependence.
* Hepatocellular disease.
* Pregnant females.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- Substance Abuse Research Center, University of Texas Health Science Center, Houston, Texas, United States